CLINICAL TRIAL: NCT05310357
Title: The Role of Chromosomal Instability in Monitoring the Course of Ovarian High-grade Serous Carcinoma
Brief Title: Chromosomal Instability in Ovarian Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Lei Li (Other)
Responsible Party: Sponsor-Investigator, Lei Li, Professor, Peking Union Medical College Hospital
Organization: Peking Union Medical College Hospital (Other)
Other Study IDs: EOC-CIN
Record Dates: First submitted 2022-03-26; First posted 2022-04-04 (Actual); Last update posted 2022-04-04 (Actual); Status verified 2022-03

CONDITIONS: Epithelial Ovarian Cancer; High-grade Serous Ovarian Carcinoma; Chromosomal Instability; Somatic Copy Number Distortion; Survival Outcomes; Minimal Residual Lesions; Progression-free Survival; Overall Survival
MeSH Terms: conditions — Carcinoma, Ovarian Epithelial; Chromosomal Instability

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — The chromosomal instability in peripheral cell-free DNA was observed before initial treatment, after primary debulking or staging surgeries, before recurrence and during the process of recurrence treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Testing for chromosomal instability (CIN) — The CIN in peripheral cell-free DNA was observed before initial treatment, after primary debulking or staging surgeries, before recurrence and during the process of recurrence treatment.

SUMMARY:
Chromosomal instability (CIN) refers to the ongoing genomic change, which involves the amplification or deletion of chromosome copy number or structure. The changes rang from point mutation to small-scale genomic change and even the change of whole chromosome number. It has been reported that the characteristics of genomic rearrangement can be used as a marker of clinical outcome of high-grade serous ovarian cancer, and specific genomic rearrangement are related to the poor prognosis. In noninvasive gene detection with low coverage, patients diagnosed with ovarian cancer have deteriorating progression-free and overall survivals regardless of the tumor stage when somatic copy number distortion (sCNA) exceeds the threshold in plasma. The detection rate of sCNA increased along with the tumor stage. We enrolled those as our target patients, who are diagnosed with high-grade serous ovarian cancer and willing to take part in. The CIN in peripheral cell-free DNA was observed before initial treatment, after primary debulking or staging surgeries, before recurrence and during the process of recurrence treatment. Our aim is to explore the application of CIN in peripheral tumor DNA in the detection of minimal residual lesions (MRD) after primary treatment and recurrence monitoring.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed of primary ovarian high grade serous carcinoma (HGSC)
* Aged 18 years or older
* Acceptance of surgical treatment for HGSC
* With detailed follow-up outcomes

Exclusion Criteria:

* Not meeting all of the inclusion criteria
* Declining to anticipate the trial

Min Age: 18 Years | Sex: Female
Age Groups: Adult, Older Adult
Study Population: Patients confirmed of primary ovarian high grade serous carcinoma.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2022-03-26 (Actual); Primary Completion 2023-03-26 (Estimated); Study Completion 2024-03-26 (Estimated)

PRIMARY OUTCOMES:
Incidence of chromosomal instability (CIN) | One year
  Incidence of chromosomal instability tested in peripheral cell-free DNA

SECONDARY OUTCOMES:
Progression-free survival | One year
  Progression-free survival in patients accepting CIN testing
Overall survival | One year
  Overall survival in patients accepting CIN testing

CONTACTS AND LOCATIONS:
Overall Officials: Lei Li, M.D., Principal Investigator — Peking Union Medical College Hospital
Locations (1):
- Lei Li, Beijing, Beijing Municipality, China